CLINICAL TRIAL: NCT02266355
Title: A Pilot Study of the Role of Omalizumab (Xolair) in Reducing the Incidence of Oxaliplatin-induced Hypersensitivity Reaction (HSR)
Brief Title: Role of Omalizumab in Reducing the Incidence of Oxaliplatin-induced Hypersensitivity Reaction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1408014510
Record Dates: First submitted 2014-10-10; First posted 2014-10-17 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Colon Cancer
Keywords: Oxaliplatin; Omalizumab
MeSH Terms: conditions — Colonic Neoplasms | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OmalizumabTreatment Group (Experimental): Omalizumab (Xolair) 300 mg SQ every 2 weeks
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab 300 mg SQ every 2 weeks
  Other Names: Xolair

SUMMARY:
Pilot study to evaluate the activity of omalizumab in the prevention of recurrent oxaliplatin hypersensitivity reaction (HSR) in oxaliplatin-sensitive patients. The study will also evaluate the safety of omalizumab (Xolair) when administered in this setting.

DETAILED DESCRIPTION:
This is an open label single arm pilot study studying the effects of omalizumab in the treatment of oxaliplatin hypersensitivity reaction (HSR) for patients with stage IV GI cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinically evident HSR to oxaliplatin, with symptoms of flushing, urticaria, pruritus, rash, and/or dyspnea without bronchospasm that emerge during or shortly after of oxaliplatin infusion
* Responding (complete or partial) or stable disease according to RECIST criteria while undergoing treatment with oxaliplatin containing regimen or need to resume an oxaliplatin based regimen in the setting of well-documented recent oxaliplatin hypersensitivity reaction
* Histologically confirmed stage IV GI cancer (AJCC 7th edition) currently sensitive to oxaliplatin containing chemotherapy regimen
* Age 18 years or older
* ECOG performance status 0-2
* Adequate bone marrow, liver, and kidney function. (WBC > 1500 cells/uL, platelets > 50,000/uL, ALT/AST < 5xULN (unless due to liver metastasis), Creatinine < 2.0 mg/ld)
* Willing to give written informed consent, adhere to the visit schedules and meet study requirements

Exclusion Criteria:

* Prior history of severe reactions to oxaliplatin as characterized by the presence of hemodynamic instability, significant respiratory symptoms or potential airway compromise
* History of hypersensitivity reaction to Xolair or any ingredient of Xolair
* Concurrent therapy with investigational agents
* Use of any other investigational agent in the last 15 days and all toxicity of prior therapy resolved
* Psychological, familial, or sociological condition potentially hampering compliance with the study protocol and follow-up schedule
* Women of childbearing potential not using the contraception method(s), as well as women who are breastfeeding
* Patients with severe medical conditions that in the view of the investigator prohibits participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence of Recurrent HSR | up to 12 months
  Recurrent Oxaliplatin HSR in subjects treated with omalizumab

SECONDARY OUTCOMES:
Safety of Omalizumab | up to 12 months
  Evaluate the safety of omalizumab by assessment of frequency of adverse events and serious adverse events as categorized by CTCAE version 4

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Stein, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States